CLINICAL TRIAL: NCT05737550
Title: A Second Explorative Pilot Study Evaluating Usability and Functionality of a New Mobile Phone Application Measuring Eye Parameters of Eyes in Patients With Confirmed Substance Use Disorder (SUD)
Brief Title: An Explorative Pilot Study of a New Mobile Phone Application Measuring Eye Parameters of Eyes in Patients With SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kontigo Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KCClin02
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The investigation aims to enroll up to 30 SUD subjects. As this is an early feasibility and explorative investigation, the sample size is not derived from a sample size calculation as no hypothesis is pre-defined. It is based on available subjects from the clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with confirmed SUD (Experimental): Evaluation of the usability of Previct Drugs when used in the intended population (patients with SUD).
  Interventions: Device: Previct Drugs

INTERVENTIONS:
Device: Previct Drugs — Previct Drugs is a new non CE-marked eHealth system intended to be used for future monitoring and treatment of patients with substance use disorder (SUD). Previct Drugs consists of an application (app) to be installed on a smartphone, a web-based careportal to be accessed from a computer by the healthcare professional for administration and access of registered data, and a database for storage, handling, and analysis of reported data. Previct Drugs is intended to be used by healthcare professionals and patients within treatment of SUD.

SUMMARY:
This will be a pre-market, explorative, early feasibility, pilot, controlled clinical investigation designed to collect initial clinical data for Previct Drugs.

DETAILED DESCRIPTION:
This second early feasibility study will give valuable information on the usability of Previct Drugs once being used in the intended population, i.e, patients with confirmed Substance Use Disorder (SUD). It will also give valuable information on the feasibility of Previct drugs function to measure pupils and eye movements in this population including evaluating the safety when using the device.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male and female
* A recurrent visitor at Sprututbytesprogrammet in Uppsala defined as visited the clinic within the last three (3) months
* SUD in accordanve with DSM-5 criteria according to investigator/designee judgement
* Age 18 and above
* Negative urine pregnancy test for all fertile women
* Been informed of the nature, the scope, and the relevance of the clinical investigation
* Voluntarily agreed on participation and has duly singed the Informed Consent Form

Exclusion Criteria:

* Participating in another clinical investigation which may affect the study outcome according to clinical judgement
* Pregnancy or lactating
* Blind
* Deaf
* Any ECG dangerous arrythmia according to the investigator or designee judgement
* Any disease or condition that may influence pupillary reflexes based on clinical judgement
* Undergone eye surgery that may influence pupillary reflexes based on clinical judgement
* Not able to read or understand the local language
* Any planned travel or treatment which will make it impossible to participate according to the investigator or designee
* Any other condition that as judged by the investigator may make the follow-up or investigation inappropriate
* That according to the Declaration of Helsinki is deemed unsuitable for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markku Hämäläinen, PhD, Study Chair — Kontigo Care AB
Locations (1):
- Mottagning för särskild vård, sprutbytet, Husläkarmottagning för hemlösa, Uppsala, Uppland, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With Confirmed SUD
Started | 24 (25 subjects signed the informed consent, out of which 24 were eligible and are included in the Full Analysis Set (FAS) population.)
Visit 2 (Follow-up Visit 1) (Optional visit) | 11 (Out of the 24 enrolled subjects, 11 (44 %) conducted the optional first follow-up visit (Visit 2).)
Visit 3 (Follow-up Visit 2) (Optional visit) | 5 (Out of the 24 enrolled subjects, 5 (20 %) conducted the optional second follow-up visit (Visit 3).)
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible subjects = Full Analysis Set (FAS)
Groups:
- Subjects With Confirmed SUD: Evaluation of the usability of Previct Drugs when used in the intended population, patients with substance use disorder (SUD).
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Timeline follow-back for drugs and alcohol. Question 1. [Count of Participants; unit: Participants] — Question 1. How often do you use drugs other than alcohol?
  * Never
  * Once a month or less often
  * 2-4 times per month
  * 2-3 times per week
  * 4 times per week or more often
  Participants
    Never | 0
    Once a month or less often | 0
    2-4 times per month | 1
    2-3 times per week | 2
    4 times per week or more often | 21
Timeline follow-back for drugs and alcohol. Question 2. [Count of Participants; unit: Participants] — Question 2. Do you use more than one drug on one occasion?
  * Never
  * Once a month or less often
  * 2-4 times per month
  * 2-3 times per week
  * 4 times per week or more often
  Participants
    Never | 4
    Once a month or less often | 1
    2-4 times per month | 5
    2-3 times per week | 2
    4 times per week or more often | 12
Timeline follow-back for drugs and alcohol. Question 3. [Count of Participants; unit: Participants] — Question 3. How many times do you take drugs during a typical day when you use drugs?
  * 0
  * 1-2 times
  * 3-4 times
  * 5-6 times
  * 7 or more
  Participants
    0 | 0
    1-2 times | 3
    3-4 times | 11
    5-6 times | 7
    7 or more | 3
Timeline follow-back for drugs and alcohol. Question 4. [Number; unit: Participants consuming the listed drug] — Question 4. What have you consumed in the last 24 hours?
  * Alcohol
  * BZ/Sleeping pills than alcohol?
  * Hashish, cannabis
  * Amphetamine, cocaine, ectasy
  * Morphine, heroine, buprenorphine, fentanyl, codeine, tramadol
  * Other
  All applicable were to be checked.
  Participants consuming the listed drug
    Alcohol | 8
    BZ/Sleeping pills than alcohol? | 10
    Hashish, cannabis | 9
    Amphetamine, cocaine, ectasy | 18
    Morphone, heroine, buprenorphine, fentanyl, codeine, tramadol | 13
    Other | 2
Timeline follow-back for drugs and alcohol. Question 5. [Count of Participants; unit: Participants] — Question 5. How affected do you feel?
  * Not affected
  * Little affected
  * Affected
  * Very affected
  Participants
    Not affected | 5
    Little affected | 18
    Affected | 1
    Very affected | 0
Timeline follow-back for drugs and alcohol. Question 6. [Count of Participants; unit: Participants] — Question 6. What has the intake looked like during the last 24 hours compared to how it usually is?
  * More than usual
  * As much as usual
  * Less than usual
  Participants
    More than usual | 4
    As much as usual | 13
    Less than usual | 7

OUTCOME MEASURES:

1. Primary Outcome: Usability Questionnaire - Question 1.
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 1. Please evaluate the study subject's ability to use the mobile phone?
  Response options:
  * Good
  * Manageable
  * Less good
Time Frame: Day 0 (Visit 1)
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  Good | 16
  Manageble | 7
  Less good | 1

2. Primary Outcome: Usability Questionnaire - Question 2
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 2. How did you perceive the study subject's ability to follow the instructions given by Previct Drugs?
  Response options:
  * Very good
  * Good
  * Either good or bad
  * Difficult
  * Very difficult
Time Frame: Day 0 (Visit 1)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  Very good | 5
  Good | 11
  Either good or bad | 6
  Difficult | 2
  Very difficult | 0

3. Primary Outcome: Usability Questionnaire - Question 4
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 4. How did the study subject experience to put him/herself in the right position to be able to start a test?
  Response options:
  * Very easy
  * Easy
  * Either easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 0 (Visit 1)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  Very easy | 2
  Easy | 12
  Either easy or difficult | 3
  Difficult | 4
  Very difficult | 3

4. Primary Outcome: Usability Questionnaire - Question 6
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 6. How would you evaluate the study subject's ability to perform a Cross-eyes test?
  Response options:
  * Very easy
  * Easy
  * Either easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 0 (Visit 1)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  Very easy | 4
  Easy | 9
  Either easy or difficult | 3
  Difficult | 6
  Very difficult | 2

5. Primary Outcome: Usability Questionnaire - Question 8
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 8. How would you evaluate the study subject's ability to perform a Nystagmus test?
  Response options:
  * Very easy
  * Easy
  * Either easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 0 (Visit 1)
Population: FAS. Analysis data missing for one subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 23
Participants
  Very easy | 10
  Easy | 7
  Either easy or difficult | 3
  Difficult | 3
  Very difficult | 0

6. Primary Outcome: Usability Questionnaire - Question 10
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 10. How would you evaluate the study subject's ability to perform a Contraction Test?
  Response options:
  * Very easy
  * Easy
  * Either easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 0 (Visit 1)
Population: FAS. Analysis data missing for one subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 23
Participants
  Very easy | 5
  Easy | 8
  Either easy or difficult | 2
  Difficult | 5
  Very difficult | 3

7. Primary Outcome: Usability Questionnaire - Question 12.
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 12. How did the study subject experience keeping the phone still during the test?
  Response options:
  * Very easy
  * Easy
  * Either easy or difficult
  * Difficult
  * Very difficult
Time Frame: Day 0 (Visit 1)
Population: FAS. Analysis data missing for one subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 23
Participants
  Very easy | 3
  Easy | 15
  Either easy or difficult | 2
  Difficult | 2
  Very difficult | 1

8. Primary Outcome: Usability Questionnaire - Question 14.
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 14. In addition to the basic instructions, did the study subject need additional support performing tests with Previct Drugs?
  Response options:
  * Yes
  * No
  * Partly
Time Frame: Day 0 (Visit 1)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  Yes | 10
  No | 14
  Partly | 0

9. Primary Outcome: Usability Questionnaire - Question 16.
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 16. Was the study subject able to perform the test after receiving additional support?
  Response options:
  * Yes
  * No
  * Partly
Time Frame: Day 0 (Visit 1)
Population: FAS, the 10 subjects answering yes to usability question 14 (secondary endpoint 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 10
Participants
  Yes | 8
  No | 1
  Partly | 1

10. Primary Outcome: Usability Questionnaire - Question 17.
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 17. How many efforts did it take the study subject to perform test with Previct Drugs?
  Response options:
  * 1-2 times
  * 3-4 times
  * More than 4 times
Time Frame: Day 0 (Visit 1)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  1-2 times | 19
  3-4 times | 4
  More than 4 times | 1

11. Primary Outcome: Usability Questionnaire - Question 18.
Description: Observation of a study subject during a test with Previct Drugs through answering a usability questionnaire consisting of 18 usability questions.
  Question 18. How likely do you think it is that the study subject will be able to perform tests with Previct Drugs without assistance in a home environment?
  Response options:
  * Very likely
  * Likely
  * Neither likely nor unlikely
  * Unlikely
  * Very unlikely
Time Frame: Day 0 (Visit 1)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Participants
  Very likely | 8
  Likely | 8
  Neither likely nor unlikely | 4
  Unlikely | 3
  Very unlikely | 1

12. Secondary Outcome: Evaluate if Self-administered Pupillometry Using a Mobile Phone Application Can be Used to Collect Pupillograms for Patients With Substance Use Disorder.
Description: The fraction of collected pupillometry data from the mobile phone application, which can be transformed into pre-defined key features using native pupillograms, i.e. proportion of successful tries. For each of the measurements pupillary light reflex (PLR), non-convergence (NC), horizontal nystagmus (NY), tremor (TR), and redness (RED) the measurements quality control will approve the measurement or not using the native pupillogram. The proportion of approved measurements over all measurements will be calculated for each of the tests (PLR, NC, NY, TR, RED). The results includes all tries performed, including tries in two ambient light conditions. In case one test is not approved by the application's quality control, the application will instruct the subject to re-do the test. The number tests are thus more than the number of subjects included in the study, and can differ between the different test types.
Time Frame: Up to 4 weeks post baseline
Population: All tries documented for each of the measurements; pupillary light reflex (PLR), non-convergence (NC), horizontal nystagmus (NY), tremor (TR), and redness (RED), for the FAS population.
Measure: Count of Units; unit: Number of tries
Units Other Than Participants: Number of tries
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Number analyzed (Number of tries) | 92
Number of tries
  Successful tries - Non-convergence (NC): number analyzed (Number of tries) | 44
  Successful tries - Non-convergence (NC) | 40
  Successful tries - Horizontal nystagmus (NY): number analyzed (Number of tries) | 41
  Successful tries - Horizontal nystagmus (NY) | 23
  Successful tries - Tremor (TR): number analyzed (Number of tries) | 41
  Successful tries - Tremor (TR) | 39
  Successful tries - Pupillary light reflex (PLR) | 79
  Successful tries - Redness (RED) | 84

13. Secondary Outcome: Evaluate if Self-administered Pupillometry Using a Mobile Phone Application, After Refinement, Can be Used to Collect Pupillograms From Patients With Substance Use Disorder.
Description: The fraction of collected pupillometry data from the mobile phone application, which can be transformed into pre-defined key features using refined pupillograms, i.e. proportion of successful tries. For each of the measurements pupillary light reflex (PLR), non-convergence (NC), horizontal nystagmus (NY), tremor (TR), and redness (RED) the measurements quality control will approve the measurement or not using the refined pupillogram. The proportion of approved measurements over all measurements will be calculated for each of the tests (PLR, NC, NY, TR, RED). The results includes all tries performed, including tries in two ambient light conditions. In case one test is not approved by the application's quality control, the application will instruct the subject to re-do the test. The number tests are thus more than the number of subjects included in the study, and can differ between the different test types.
Time Frame: Up to 4 weeks post baseline
Population: as for outcome 12
Measure: Count of Units; unit: Number of tries
Units Other Than Participants: Number of tries
Arm/Group | Subjects With Confirmed SUD
Number analyzed (Participants) | 24
Number analyzed (Number of tries) | 92
Number of tries
  Successful tries - Non-convergence (NC): number analyzed (Number of tries) | 44
  Successful tries - Non-convergence (NC) | 40
  Successful tries - Horizontal nystagmus (NY): number analyzed (Number of tries) | 41
  Successful tries - Horizontal nystagmus (NY) | 23
  Successful tries - Tremor (TR): number analyzed (Number of tries) | 41
  Successful tries - Tremor (TR) | 39
  Successful tries - Pupillary light reflex (PLR) | 79
  Successful tries - Redness (RED) | 84

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 weeks.
Arm/Group | Subjects With Confirmed SUD
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT05737550/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT05737550/SAP_001.pdf